CLINICAL TRIAL: NCT04888234
Title: Evaluation the Effectiveness of Ru-Yi-Jin-Huang Powder for the Radiation-induced Dermatitis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202000655A3
Record Dates: First submitted 2021-05-10; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Radiation Dermatitis
Keywords: Radiation dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The treatment group receive topical treatment of Ru-Yi-Jin-Huang Powder.
  Interventions: Drug: Ru-Yi-Jin-Huang Powder
- Control group (No Intervention): The control group receive regular management for radiation-induced dermatitis.

INTERVENTIONS:
Drug: Ru-Yi-Jin-Huang Powder — Ru-Yi-Jin-Huang Powder is the most common TCM topical drug for skin diseases. It is often used to treat skin ulcers, sprain of joint with swelling, and other inflammatory diseases.
  Arms: Treatment group

SUMMARY:
Radiation-induced dermatitis is the most common complication of radiotherapy for cancer treatment. However, there is no satisfactory management to deal with the problem. Ru-Yi-Jin-Huang Powder is one of most common topical TCM drug to treat skin diseases but lack of evidence to support efficacy. The aim of this trial is to evaluate the effectiveness of Ru-Yi-Jin-Huang Powder for radiation-induced dermatitis.

DETAILED DESCRIPTION:
The common management of head and neck cancer are concurrent chemoradiotherapy (CCRT) after surgical section. Radiation-induced dermatitis is the most common complication of radiotherapy for cancer, affecting approximately 95 percent of patients receiving radiotherapy. The skin changes include erythema, edema, pigment changes, hair loss, and dry or moist desquamation. It may cause xerostomia, hard food taking, severe infection to delay the completion of course of treatment. Although, there are lots of topical drug to deal with radiation dermatitis, there is no best way to manage the skin problems. Ru-Yi-Jin-Huang Powder is one of most common topical TCM drug to treat skin ulcer, joint swelling or other infective or inflammatory diseases. Some study showed that Ru-Yi-Jin-Huang Powder can be used to decrease edema or swelling, pain relief, decrease phlebitis or mumps. However, there is no related evidence to support Ru-Yi-Jin-Huang Powder for radiation dermatitis. Thus, the aim of the study is to evaluate the effectiveness of Ru-Yi-Jin-Huang Powder for radiation-induced dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* stage 3 or 4 of head and neck cancer or nasopharyngeal cancer with pathological confirmed malignancy undergoing concurrent chemoradiotherapy more than 20 times or radiation dermatitis > CTCAE grade 2.
* more than 18 years old.
* VAS score > 6 with poor response to narcotics.
* estimated survival time of > 6 months.
* be suitable for TCM topical treatment after evaluation by TCM physicians.
* willingness to joint this trial and sign consent form of study.

Exclusion Criteria:

* non-head and neck cancer or have not receive CCRT.
* not be suitable for Ru-Yi-Jin-Huang topical treatment after TCM physicians evaluation.
* history of allergy to TCM topical use.
* poor conscious to answer questionnaires.
* pregnancy.
* KPS < 30.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-08 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Change of VAS score from baseline and 2 months | VAS score is assessed by physicians 2 times a week, up to 8 weeks.
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 0 of 'no pain at all' and 10 of 'pain as bad as it could be'.
Change of CTCAE version 4 from baseline and 2 months | CTCAE is assessed by physicians once a week with photos following, up to 8 weeks.
  The criteria is used for the management of chemoradiotherapy administration. and dosing, and to provide standardization and consistency in the definition of treatment-related toxicity.
Change of Skindex-16 from baseline and 2 months | Skindex-16 is assessed by physicians once a week, up to 8 weeks.
  The scale is a brief quality-of-life measure for patients with skin diseases.